CLINICAL TRIAL: NCT02653287
Title: Lupus Intervention for Fatigue Trial
Acronym: LIFT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Rosalind Ramsey-Goldman, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LIFT Study
Record Dates: First submitted 2016-01-07; First posted 2016-01-12 (Estimated); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Fatigue; Physical Activity; Lupus Erythematosus, Systemic
Keywords: Fatigue, Physical Activity, Lupus
MeSH Terms: conditions — Fatigue; Motor Activity; Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The experimental intervention is a unique combination of four individual counseling sessions based in motivational interviewing focusing on physical activity, dietary behavior and behavioral strategies. The individual sessions will provide a tailored personalized intervention including problem-solving and goal setting for increasing physical activity, and following a healthy diet. Healthy Lifestyle Coaches (RN or MPH) will be responsible for conducting the individual for a caseload of participants. There are no drugs involved in the intervention.
  Interventions: Behavioral: Experimental
- Control (Active Comparator): The control group intervention will receive four individual phone calls checking in with participants regarding questions about the study or from the educational sessions focusing on SLE disease management, each lasting approximately 10-15 minutes.
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Experimental — The experimental intervention includes 4 individual coaching sessions (initial 1 hour in-person and remaining 10-15 minutes per telephone) designed to identify barriers and supports for physical activity and nutrition using motivational interviewing. They occur shortly after randomization, 1.5, 3, and 6 months. Daily participants monitor their physical activity via the Fitbit Flex and their dietary behavior on a paper diary.
  Arms: Intervention
Other: Control — The control group will receive four individual phone calls focusing on education for SLE disease management, as well as answering any questions the participants have about the study. Topics include: what is lupus, laboratory tests, medications, taking charge of your health care and managing stress (2 sessions). Each call will last about 10-15 minutes, and occur shortly after randomization, then at 1.5, 3, and 6 months.
  Arms: Control

SUMMARY:
Participants in the Chicago Lupus Database or individuals seen at Northwestern Medicine will be approached to enroll in a one year clinical trial looking at decreasing fatigue in persons with systemic lupus erythematosus (SLE). The intervention group will receive individual coaching sessions focusing on physical activity and nutrition while the control group will receive individual calls in relation to SLE self-management educational sessions.This study is designed to evaluate the LIFT intervention to decrease fatigue (primary outcome), improve physical activity (secondary outcome) and dietary behavior (exploratory outcome) in persons with SLE.

DETAILED DESCRIPTION:
Participants in the Chicago Lupus Database or individuals seen at Northwestern Medicine will be approached to enroll in a one year clinical trial looking at decreasing fatigue in persons with systemic lupus erythematosus (SLE). The intervention group will receive individual coaching based in motivational interviewing sessions focusing on physical activity and nutrition while the control group will receive individual calls focusing on SLE self-management. This study is designed to evaluate the LIFT intervention to decreased fatigue (primary outcome), improve physical activity (secondary outcome) and dietary behavior (exploratory outcome) in persons with SLE.

ELIGIBILITY:
Inclusion criteria:

* include meeting at least 4 of 11 American College of Rheumatology (ACR) classification criteria for definite SLE, or 3 out of 11 ACR classification criteria with also meeting at least one SLICC criteria
* be at least 18 years of age
* have a BMI between 18-40 kg/m2
* be able to ambulate at least household distances (50ft)
* be able to provide informed consent.
* be able to speak and read English

Exclusion criteria:

* include pregnancy at baseline
* not meeting inclusion criteria.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Fatigue Severity Scale over time | Baseline, 3, 6, 12 months
  Online questionnaire

SECONDARY OUTCOMES:
Change in Physical Activity Scale over time | Baseline, 3, 6, 12 months
  Accelerometry
Change in International Physical Activity Questionnaire (IPAQ) over time | Baseline, 3, 6, 12 months
  Phone Interview Questionnaire
Godin Leisure Time Exercise Questionnaire | Baseline, 6, 12 months
  Phone Interview Questionnaire

OTHER OUTCOMES:
Change in Nutrition Data Systems for Research (NDSR) over time | Baseline, 6, 12 months
  Dietary Recall Interview

CONTACTS AND LOCATIONS:
Overall Officials: Rosalind Ramsey-Goldman, MD, DrPH, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Holly Milaeger, Chicago, Illinois
  - Northwestern University, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: Yes
It is the intent of all investigators in this project to share any and all resources generated as a result of an award for this project. The final data from this project will be de-identified in accordance with HIPAA guidelines.

REFERENCES:
- [Background] Ramsey-Goldman R, Rothrock N. Fatigue in systemic lupus erythematosus and rheumatoid arthritis. PM R. 2010 May;2(5):384-92. doi: 10.1016/j.pmrj.2010.03.026. PMID 20656619
- [Background] del Pino-Sedeno T, Trujillo-Martin MM, Ruiz-Irastorza G, Cuellar-Pompa L, de Pascual-Medina AM, Serrano-Aguilar P; Spanish Systemic Lupus Erythematosus CPG Development Group. Effectiveness of Nonpharmacologic Interventions for Decreasing Fatigue in Adults With Systemic Lupus Erythematosus: A Systematic Review. Arthritis Care Res (Hoboken). 2016 Jan;68(1):141-8. doi: 10.1002/acr.22675. PMID 26238554
- [Background] Ahn GE, Chmiel JS, Dunlop DD, Helenowski IB, Semanik PA, Song J, Ainsworth B, Chang RW, Ramsey-Goldman R. Self-reported and objectively measured physical activity in adults with systemic lupus erythematosus. Arthritis Care Res (Hoboken). 2015 May;67(5):701-7. doi: 10.1002/acr.22480. PMID 25251755
- [Background] Mancuso CA, Perna M, Sargent AB, Salmon JE. Perceptions and measurements of physical activity in patients with systemic lupus erythematosus. Lupus. 2011 Mar;20(3):231-42. doi: 10.1177/0961203310383737. Epub 2010 Dec 23. PMID 21183562
- [Background] Ramsey-Goldman R, Schilling EM, Dunlop D, Langman C, Greenland P, Thomas RJ, Chang RW. A pilot study on the effects of exercise in patients with systemic lupus erythematosus. Arthritis Care Res. 2000 Oct;13(5):262-9. doi: 10.1002/1529-0131(200010)13:53.0.co;2-8. PMID 14635294
- [Background] Davies RJ, Lomer MC, Yeo SI, Avloniti K, Sangle SR, D'Cruz DP. Weight loss and improvements in fatigue in systemic lupus erythematosus: a controlled trial of a low glycaemic index diet versus a calorie restricted diet in patients treated with corticosteroids. Lupus. 2012 May;21(6):649-55. doi: 10.1177/0961203312436854. Epub 2012 Feb 6. PMID 22311939
- [Background] Lin JS, O'Connor E, Whitlock EP, Beil TL. Behavioral counseling to promote physical activity and a healthful diet to prevent cardiovascular disease in adults: a systematic review for the U.S. Preventive Services Task Force. Ann Intern Med. 2010 Dec 7;153(11):736-50. doi: 10.7326/0003-4819-153-11-201012070-00007. PMID 21135297
- [Background] Delahanty LM. Research charting a course for evidence-based clinical dietetic practice in diabetes. J Hum Nutr Diet. 2010 Aug;23(4):360-70. doi: 10.1111/j.1365-277X.2010.01065.x. Epub 2010 Apr 27. PMID 20456590
- [Background] Krupp LB, LaRocca NG, Muir-Nash J, Steinberg AD. The fatigue severity scale. Application to patients with multiple sclerosis and systemic lupus erythematosus. Arch Neurol. 1989 Oct;46(10):1121-3. doi: 10.1001/archneur.1989.00520460115022. PMID 2803071